CLINICAL TRIAL: NCT05778695
Title: Brain Small Chain Fatty Acid Metabolism in Parkinson Disease: Ketones
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawal of funding
Sponsor: University of Michigan (Other)
Collaborators: Farmer Family Foundation (Unknown)
Responsible Party: Principal Investigator, Nicolaas Bohnen, MD, PhD, Professor, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00213035
Record Dates: First submitted 2023-02-21; First posted 2023-03-21 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; Lewy Body Dementia; Parkinson Disease Dementia
Keywords: ketone ester; ketosis; functional neuroimaging
MeSH Terms: conditions — Parkinson Disease; Lewy Body Disease; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parkinson Disease (Experimental): Participants will take the ketone ester supplement for 30 days +/- 7 days. For days 1 through 7, participants will take 12.5g (25mL) of the ketone ester supplement (KetoneAid) TID, and on day 8, the dose will be increased to 25g (50mL) three times daily (TID) as tolerated. KE dose will be titrated down to a tolerated level if necessary.
  Interventions: Dietary Supplement: Ketone Ester (R)-3-Hydroxybutyl (R)-3-Hydroxybutyrate
- Parkinson Disease Dementia/Lewy Body Dementia (Experimental): Participants will take the ketone ester supplement for 30 days +/- 7 days. For days 1 through 7, participants will take 12.5g (25mL) of the ketone ester supplement (KetoneAid) TID, and on day 8, the dose will be increased to 25g (50mL) TID as tolerated. KE dose will be titrated down to a tolerated level if necessary.
  Interventions: Dietary Supplement: Ketone Ester (R)-3-Hydroxybutyl (R)-3-Hydroxybutyrate
- Healthy Controls (Experimental): Participants will take the ketone ester supplement for 30 days +/- 7 days. For days 1 through 7, participants will take 12.5g (25mL) of the ketone ester supplement (KetoneAid) TID, and on day 8, the dose will be increased to 25g (50mL) TID as tolerated. KE dose will be titrated down to a tolerated level if necessary.
  Interventions: Dietary Supplement: Ketone Ester (R)-3-Hydroxybutyl (R)-3-Hydroxybutyrate

INTERVENTIONS:
Dietary Supplement: Ketone Ester (R)-3-Hydroxybutyl (R)-3-Hydroxybutyrate — Ketone ester (KE) dietary supplement (KetoneAid)
  Other Names: KetoneAid

SUMMARY:
Small exploratory open-label pilot study to assess supplementation of a ketone ester (KetoneAid) as a potential therapy for persons with Parkinson disease (PD), Parkinson Disease Dementia/Lewy Body Dementia (PDD/LBD), and healthy controls.

DETAILED DESCRIPTION:
The overarching goal of this study is to investigate glucose metabolic, cognitive, clinical and imaging changes in persons with PD and PDD/LBD before and after a month supplementation of a ketone ester (KetoneAid) in a small open label exploratory clinical trial. Positive findings in this small exploratory pilot trial may support future target engagement studies of ketone supplementation in PD and normal adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control volunteers over 45 years of age
* People with Parkinson Disease over 45 years of age
* People with Parkinson's Disease Dementia or Lewy Body Dementia over 45 years of age

Exclusion Criteria:

* Participants with contra-indications to MR imaging, including pacemakers or claustrophobia;
* Evidence of large vessel stroke or mass lesion on MRI
* Regular use of anti-cholinergic, benzodiazepines, high dose (>100mg QD) of quetiapine, or neuroleptic drugs
* History of significant GI disease
* Significant metabolic or uncontrolled medical comorbidity
* Poorly controlled diabetes
* Pregnancy or breast feeding
* Current excessive alcohol use
* Suicidal ideation

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas Bohnen, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Domino's Farms, Ann Arbor, Michigan
  - University Hospital, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 participants were enrolled in the study. There were no withdrawals.
Period: Overall Study
Arm/Group | Parkinson Disease | Parkinson Disease Dementia/Lewy Body Dementia | Healthy Controls
Started | 4 | 10 | 2
Completed | 4 | 10 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parkinson Disease | Parkinson Disease Dementia/Lewy Body Dementia | Healthy Controls | Total
Number analyzed (Participants) | 4 | 10 | 2 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 4 | 10 | 2 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 77 (4.03) | 74.5 (4.93) | 70 (1.41) | 74.63 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 2 | 10 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 10 | 2 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 10 | 2 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 10 | 2 | 16
Education [Mean (Standard Deviation); unit: years] | 19.0 (3.56) | 16.7 (4.52) | 17.0 (1.41) | 17.31 (4.00)
Modified Unified Parkinson's Disease Rating Scale Part 3 (MDS-UPDRSIII) [Mean (Standard Deviation); unit: units on a scale] — The Modified Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part 3 is a clinician-administered motor exam consisting of 18 items to evaluate the motor symptom severity in Parkinson's disease. Total scores range from 0 to 132, with higher scores indicating higher severity of motor symptoms. MDS-UPDRS Part 3 scores of 32 and below are typically considered mild, 33-58 is moderate, and 59 and above considered severe.
  units on a scale | 46.00 (5.90) | 47.80 (11.22) | 6.75 (9.55) | 44.23 (16.76)
Montreal Cognitive Assessment (MoCA) [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is used for detection of mild cognitive impairment. It assesses short-term memory, visuospatial abilities, executive functioning, attention, language, and orientation. Scores range from 0 to 30, with low scores indicating more cognitive impairment. Scores of 26 and above indicate normal cognitive performance, 18-25 indicate mild impairment, 10-17 indicate moderate impairment, and 0-9 indicate severe impairment.
  units on a scale | 22.25 (4.27) | 17.00 (7.41) | 24.00 (1.41) | 19.19 (6.75)
Parkinson's Disease Cognitive Rating Scale (PDCRS) [Mean (Standard Deviation); unit: units on a scale] — The Parkinson's Disease Cognitive Rating Scale (PDCRS) evaluates cognition in Parkinson's disease. Scores range from 0-134 with lower scores indicating increased cognitive impairment.
  units on a scale | 66.75 (16.13) | 48.50 (25.31) | 79.00 (7.07) | 56.88 (24.04)

OUTCOME MEASURES:

1. Primary Outcome: Glucose Metabolism
Description: Continuous glucose meter 7-10-day average glucose readings before/after open-label treatment with the ketone ester in patients with PD, Parkinson's disease dementia/Lewy body dementia, and normal controls. Healthy fasting blood glucose ranges from 70 to 99 milligrams per deciliter (mg/dL), with a healthy maximum of 180 mg/dL within 2 hours of eating meals.
Time Frame: Pre and post approximately 30 days of intervention
Population: 13 of the 16 participants completed continuous glucose monitoring. The remaining 3 participants did not complete continuous glucose monitoring due to device availability and ability to understand instructions. Healthy control sample size (n=2) was not sufficient to perform statistical analysis for that group.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Groups:
- Parkinson Disease Dementia/Lewy Body Dementia; Healthy Controls: Participants will take the ketone ester supplement for 30 days +/- 7 days. For days 1 through 7, participants will take 12.5g (25mL) of the ketone ester supplement (KetoneAid) TID, and on day 8, the dose will be increased to 25g (50mL) three times daily (TID) as tolerated. KE dose will be titrated down to a tolerated level if necessary.
  Ketone Ester (R)-3-Hydroxybutyl (R)-3-Hydroxybutyrate: Ketone ester (KE) dietary supplement (KetoneAid)
Arm/Group | Parkinson Disease | Parkinson Disease Dementia/Lewy Body Dementia | Healthy Controls
Number analyzed (Participants) | 4 | 7 | 2
milligrams per deciliter (mg/dL)
  Pre-intervention | 133.0 (20.30) | 134.86 (24.30) | 179.50 (19.09)
  Post-intervention | 128.25 (18.26) | 132.86 (33.42) | 170.50 (21.92)
Statistical Analysis 1: Comparison: Parkinson Disease; Test type: Other — A comparison is not being made between two different treatment groups. Exploratory analysis; p = 0.875, Wilcoxon (Mann-Whitney) — A priori threshold for statistical significance is p < 0.05; Median Difference (Net) = -14, Standard Deviation 22.02
Statistical Analysis 2: Comparison: Parkinson Disease Dementia/Lewy Body Dementia; Test type: Other — A comparison is not being made between two different treatment groups. Exploratory analysis; p = 0.739, t-test, 2 sided — A priori threshold for statistical significance is p < 0.05; Mean Difference (Net) = -2, 95% CI 2-sided [-16.026 to 12.026], Standard Deviation 15.166

2. Primary Outcome: Clinical Dementia Rating Scale Score
Description: The clinical dementia rating scale is a measure of functional and cognitive performance relevant to dementia. It is scored from 0 (normal) to 3 (severe dementia). The clinical dementia rating scale will be assessed in patients with Parkinson's disease, Parkinson's disease dementia/Lewy body dementia, and healthy controls before and after open-label treatment with the ketone ester.
Time Frame: Pre and post approximately 30 days of intervention
Population: All participants completed CDR before and after intervention. There was no change in CDR scores in the Parkinson's disease group, and the Healthy Control group had insufficient sample size (n = 2) to perform any statistical analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Parkinson Disease Dementia/Lewy Body Dimentia; Healthy Controls: Participants will take the ketone ester supplement for 30 days +/- 7 days. For days 1 through 7, participants will take 12.5g (25mL) of the ketone ester supplement (KetoneAid) TID, and on day 8, the dose will be increased to 25g (50mL) three times daily (TID) as tolerated. KE dose will be titrated down to a tolerated level if necessary.
  Ketone Ester (R)-3-Hydroxybutyl (R)-3-Hydroxybutyrate: Ketone ester (KE) dietary supplement (KetoneAid)
Arm/Group | Parkinson Disease | Parkinson Disease Dementia/Lewy Body Dimentia | Healthy Controls
Number analyzed (Participants) | 4 | 10 | 2
score on a scale
  Pre-intervention | 0.5 (0.41) | 1.0 (0.85) | 0 (0)
  Post-intervention | 0.5 (0.41) | 1.15 (0.88) | 0.25 (0.35)
Statistical Analysis 1: Comparison: Parkinson Disease Dementia/Lewy Body Dimentia; Test type: Other — A comparison is not being made between two different treatment groups. Exploratory analysis; p = 0.37, Wilcoxon (Mann-Whitney) — A priori threshold for statistical significance is p < 0.05; Median Difference (Net) = 0, Standard Deviation 0.34

ADVERSE EVENTS:
Time Frame: For all subjects, data was collected during the 30 +/- 7 days of tributyrin intervention.
Arm/Group | Parkinson Disease | Parkinson Disease Dementia/Lewy Body Dementia | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/10 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/10 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 8/10 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parkinson Disease (N=4) | Parkinson Disease Dementia/Lewy Body Dementia (N=10) | Healthy Controls (N=2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated, unexpected AE
Ear Infection (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) — Unrelated, unexpected AE
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Unrelated, unexpected AE
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Possibly related, expected AE
Freezing of Gait (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated, unexpected AE
Diarrhea (Gastrointestinal disorders) | 1 (2) | 2 (2) | 1 (1) — Possibly related, expected AE
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated, unexpected AE
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) — Possibly related, expected AE
Heartburn (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) — Possibly related, expected AE
Lightheadedness (Metabolism and nutrition disorders) | 2 (2) | 4 (7) | 0 (0) — Possibly related, expected AE
Low energy (General disorders) | 1 (1) | 0 (0) | 0 (0) — Unrelated, unexpected AE
Low glucose (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Possibly related, expected AE
Discomfort in Scanner (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) — Related, expected AE
Sleep changes (General disorders) | 1 (1) | 0 (0) | 0 (0) — Possibly related, expected AE
Muscle soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Possibly related, expected AE
Stomach ache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Possibly related, expected AE
Throat irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) — Possibly related, expected AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT05778695/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT05778695/ICF_000.pdf